CLINICAL TRIAL: NCT04923490
Title: Evaluation of State and Trait Anxiety Levels in Adolescents Undergoing Endoscopy Under Anesthesia
Brief Title: Anxiety Levels in Adolescents Undergoing Endoscopy
Status: Completed | Type: Observational
Sponsor: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Umran Karaca, Principal investigator, Bursa Yuksek Ihtisas Training and Research Hospital
Other Study IDs: bursa hospital
Record Dates: First submitted 2021-06-03; First posted 2021-06-11 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Anxiety
Keywords: Adolescent; anxiety; endoscopy; anesthesia
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: state and trait anxiety scale levels — While the STAI-I anxiety level is scored as "(1) never, (2) somewhat, (3) frequently, and (4) almost always", the scoring options in STAI-II are "(1) almost never, (2) sometimes, (3) most of the time, and (4) almost always".

SUMMARY:
The aim of our study was to evaluate the pre-procedure state and trait anxiety levels of adolescents patients hospitalized for the purpose of gastrointestinal endoscopy performed under sedation.

DETAILED DESCRIPTION:
Although anxiety is known to be a disorder that is much more relevant for adults, it is seen at a frequency of approximately 6.5% in the childhood and adolescence. Anxiety is usually examined in two different forms, state anxiety and trait anxiety. A total of 180 pediatric patients who underwent GIS endoscopy in our hospital were included in our study. Demographic data (age, gender, height, weight, educational status, school and grade), additional diseases and diagnoses were recorded. Our aim was to evaluate the anxiety and trait anxiety levels of adolescents scheduled for gastrointestinal system (GIS) endoscopy under sedation, after being admitted as a single-day inpatient and before the procedure. A form evaluating state and trait anxiety levels (Spielberger's state and trait anxiety scale) and another form consisting of demographic data were given to the patients. We requested that the forms be filled by the children themselves. After monitoring in the endoscopy unit, sedation was applied with IV anesthetic drugs routinely.Oxygenation was provided with nasal O2 in all patients. Heart rate (HR), mean arterial pressure (MAP) and oxygen saturation (SpO2) were monitored. Also complications (bradycardia, tachycardia, arrhythmia, hypotension, hypertension, bronchospasm, decrease in SpO2, apnea) were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 11-18 years
* ASA I-II
* cooperative
* literate
* undergoing elective endoscopic procedures

Exclusion Criteria:

* under 11 years of age
* uncooperative
* illiterate
* had known psychiatric disorders or were using psychiatric drugs
* emergency endoscopy

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 180 pediatric patients
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
anxiety level | before anesthesia induction
  Score between 0-19: No anxiety Score between 20-39: Mild anxiety Score between 40-59: Moderate anxiety Score between 60-79: Severe anxiety 80 and above score: Panic level anxiety

CONTACTS AND LOCATIONS:
Overall Officials: Ümran Ü Karaca, MD, Principal Investigator — Bursa Yuksek Ihtisas Training and Research Hospital; Derya D Karasu, Assoc Prof, Study Chair — Bursa Yuksek Ihtisas Training and Research Hospital; Şermin Ş Eminoğlu, MD, Study Chair — Bursa Yuksek Ihtisas Training and Research Hospital; Şeyda Efsun ŞE Özgünay, Assoc Prof, Study Chair — Bursa Yuksek Ihtisas Training and Research Hospital; Tuğba T Onur, MD, Study Chair — Bursa Yuksek Ihtisas Training and Research Hospital
Locations (1):
- Bursa YIERH, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Abstract of record